CLINICAL TRIAL: NCT03599856
Title: TraceBook: the Clinical Proof of Concept on the Intensive Care.
Acronym: TraceBook
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Eindhoven University of Technology (Other); Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Principal Investigator, Ashley De Bie, Physician-scientist, Catharina Ziekenhuis Eindhoven
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: nWMO-2018.61
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Critical Illness; Safety Issues
Keywords: Checklist; Intensive Care Unit; Clinical decision support systems; Medical errors; Patient safety
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: A prospective single center (Catharina Hospital Eindhoven) controlled before-and-after study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Before" control group (No Intervention): Control group with observation of current local standard of care with paper checklist available at the bedside during the ICU rounds of the ICU physicians (as usual)
- "After" Intervention group (Experimental): An mini Ipad providing TraceBook' intelligent dynamic clinical checklists during the ICU rounds of the ICU physicians.
  Interventions: Other: TraceBook

INTERVENTIONS:
Other: TraceBook — TraceBook offers the user intelligent dynamic clinical checklist that shows patient specific items to a specific user while being context aware.
  Other Names: Dynamic clinical checklist
  Arms: "After" Intervention group

SUMMARY:
The effectiveness of current checklists is hampered by lack of acceptance and compliance. Recently, a new type of checklist with dynamic properties has been created to provide more specific checklist items for each individual patient. The proof of concept of this dynamic clinical checklist (DCC; BJA 2017 (DOI: 10.1093/bja/aex129)) was tested in a simulation trial with improved outcomes and high acceptance scores. The purpose of this study is to investigate if the outcomes of this real-life clinical proof of concept study are similar with the outcomes of the simulation trial for the intensive care unit (ICU) ward.

DETAILED DESCRIPTION:
Method A prospective single center (Catharina Hospital Eindhoven) controlled before-and-after study.

The before period will be used as control group in which ward rounds and nurse handovers will be observed by the investigators for two months. Then TraceBook will be introduced and clinicians, ICU doctors and nurses, will be able to use checklists of TraceBook for ward rounds, their shifts and handovers in which they will be observed for two months. The goal is at least 120 observations per period.

Endpoints The primary outcome is the percentage of items that were checked per ward rounds and nurse handovers during the before and the after implementation period. Secondary outcomes will be clinical outcomes of admitted patients, pharmacist specific outcomes, specific checkable item related outcomes, and user experience and acceptance scores.

Hypothesis TraceBook, with the use of digital dynamic checklists, improves compliance to care processes on the intensive care with a high user acceptance score.

ELIGIBILITY:
Inclusion Criteria:

* Physicians working on the ICU
* All admitted patients on the ICU during the study periods.

Exclusion Criteria:

* Physicians objecting participation in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2019-02-12 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Checked items | 24 hours (each day)
  The percentage of daily checked checkable items overall and items requiring an intervention per patient.

SECONDARY OUTCOMES:
Mortality | 9 months
  Intensive Care mortality
Mortality | 9 months
  30 day mortality
Mortality | 9 months
  90 day mortality
Length of stay | 9 months
  Length of stay at the intensive care
Ventilator days | 9 months
  Number of days with use of mechanical ventilator (per patient and overall per period)
Sedation days | 9 months
  Number of patient days with a Richmond Agitation-Sedation Scale (score -5 till +4) between -5 and -1 as worse outcome.
Daily intensive care medication alerts | 4 months
  Number of daily intensive care medication alerts for the pharmacist.
Pharmacists' interventions | 4 months
  Types of pharmacists' interventions based on the daily intensive care medication alerts
Number of gastro-intestinal bleedings | 4 months
  The number of patients during each period with hematemesis or melena, not being the reason of admission.
Ventilator and hospital associated pneumonia on the intensive care. | 4 months
  The number of patients during each period with ventilator and hospital associated pneumonia, not being the reason of admission.
Central-venous-catheter-related bloodstream infections. | 4 months
  The number of patients during each period with central-venous-catheter-related bloodstream infections, not being the reason of admission.
Incorrect prescribed anticoagulation or thrombosis prophylaxis. | 4 months
  Number of patient days where anticoagulation or thrombosis prophylaxis is prescribed incorrect based on local protocol.
Incorrect prescribed proton pump inhibitors | 4 months
  Number of patient days where proton pump inhibitors are prescribed incorrect based on local protocol.
Incorrect prescribed selective digestive decontamination | 4 months
  Number of patient days where selective digestive decontamination is prescribed incorrect based on local protocol.
Spontaneous breathing trials | 4 months
  Number of spontaneous breathing trials when required based on local protocol in weaning patients
Sedation wake up calls | 4 months
  Number of sedation wake up calls when required based on local protocol
Intravenous sedatives use | 4 months
  Number of patient days with the use of intravenous sedatives (eg Propofol, Midazolam)
Opiates use | 4 months
  Number of patient days with the use of opiates overall and in patients with low Visual Analogue Scale scores (<4).
Antibiotics use | 4 months
  Number of patient days with the use of antibiotics overall and when not required based on local protocol.
Complication registration | 4 months
  Number of complications that were discussed within 24hrs and registered.
Energy deficit | 4 months
  Number of patient days with energy deficit of >250.
Automatically checked items | 4 months
  Number of items that where or could have been checked automatically during each period.
User experience outcomes | 6 months
  Attrakdiff questionnaire after both periods Technology Acceptance Model 2 (TAM2) based questionnaire Semi-structured interview
Hedonic and pragmatic quality | 6 months
  Attrakdiff questionnaire
User acceptance | 6 months
  Technology Acceptance Model 2 (TAM2) based questionnaire after both periods to compare paper checklist and electronic health records with digital checklist and electronic health records.
User experience | 6 months
  Semi-structured interview after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Korsten, Prof MD, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD is available if researchers ask for it.

REFERENCES:
- [Result] De Bie AJR, Nan S, Vermeulen LRE, Van Gorp PME, Bouwman RA, Bindels AJGH, Korsten HHM. Intelligent dynamic clinical checklists improved checklist compliance in the intensive care unit. Br J Anaesth. 2017 Aug 1;119(2):231-238. doi: 10.1093/bja/aex129. PMID 28854530
- [Derived] De Bie AJR, Mestrom E, Compagner W, Nan S, van Genugten L, Dellimore K, Eerden J, van Leeuwen S, van de Pol H, Schuling F, Lu X, Bindels AJGH, Bouwman ARA, Korsten EHHM. Intelligent checklists improve checklist compliance in the intensive care unit: a prospective before-and-after mixed-method study. Br J Anaesth. 2021 Feb;126(2):404-414. doi: 10.1016/j.bja.2020.09.044. Epub 2020 Nov 17. PMID 33213832

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03599856/Prot_SAP_000.pdf